CLINICAL TRIAL: NCT03733743
Title: Day-night Rhythm in Muscle Metabolism of Prediabetic Subjects
Brief Title: Day-night Rhythm in Muscle Metabolism of Prediabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL64753.068.18
Record Dates: First submitted 2018-09-19; First posted 2018-11-07 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2018-09

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Resistance
Keywords: Circadian Rhythm
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Standardized living protocol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standardized living protocol (Other): Subjects are kept at the research facility to adhere to a standardized living protocol, mimicking a normal daily living situation. During the study, multiple tests will be performed, including muscle biopsies, blood draws, MRS measurements and indirect calorimetry.
  Interventions: Other: Standardized living protocol

INTERVENTIONS:
Other: Standardized living protocol — Subjects stay at the research facility for 44 hours and adhere to a standard sleeping, eating and activity protocol. During this protocol, multiple measurements will be performed including skeletal muscle biopsies (m. vastus lateralis), blood draws, indirect calorimetry and MRS measurements.

SUMMARY:
This study evaluates the existence of a day-night rhythm in skeletal muscle energy metabolism in prediabetic subjects. Subjects will stay at the research facility for 44 hours with a standardized living protocol during which several measurements of skeletal muscle and whole body energy metabolism will be performed.

DETAILED DESCRIPTION:
Recent evidence from both observational and experimental studies indicates that disobedience of a normal day-night rhythm negatively influences metabolic and cardiovascular health, possibly leading to obesity and type 2 diabetes mellitus (T2DM). An important hallmark of obesity and T2DM is a decreased skeletal muscle mitochondrial function. Interestingly, recent research indicates that also skeletal muscle mitochondrial function is under the influence of a day-night rhythm. In this study, the presence of a day-night rhythm in skeletal muscle energy metabolism (in particular mitochondrial function) of overweight prediabetic participants will be investigated. During this study, subjects will stay at the research unit for 44 hours, with standardized meals and sleeping time. Five muscle biopsies (v. lateralis) and frequent blood draws will be taken. In addition, indirect calorimetry measurements will be performed.

ELIGIBILITY:
Inclusion criteria:

* Caucasian
* Healthy (as determined by dependent physician)
* Overweight: BMI 25 - 35 kg/m2
* Prediabetic based on one or a combination of the following criteria:

  * Impaired Glucose Tolerance (IGT): plasma glucose values ≥ 7.8 mmol/l and ≤ 11.1 mmol/l 120 minutes after glucose drink consumption during OGTT in screening.
  * Impaired Fasting Glucose (IFG): Fasting plasma glucose ≥ 6.1 mmol/l and ≤ 6.9 mmol/l.
  * Insulin Resistance: glucose clearance rate ≤ 360ml/kg/min, as determined using the OGIS120 model.
  * HbA1c of 5.7-6.4%.
* Regular sleeping time (normally 7 - 9h daily)
* Stable dietary habits: no weight gain or loss > 3kg in the last three months.

Exclusion criteria:

* Use of anticoagulants
* Previously diagnosed with type 2 diabetes
* Current alcohol consumption > 20 grams alcohol/day
* Extreme early bird or extreme night person (score ≤ 30 or ≥ 70 on MEQ-SA questionnaire)
* Heavily varying sleep-wake rhythm
* Nightshift work during last 3 months
* Travel across > 1 time zone in the last 3 months
* Significant food allergies/intolerance (seriously hampering study meals)
* Using > 400mg caffeine daily (more than 4 coffee or energy drink)
* Smoking

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Day-night rhythm in skeletal muscle mitochondrial respiration | measured on day two at 8:00, 13:00, 18:00, 23:00, 04:00
  O2-flux (pmol/mg/s) measured with high resolution respirometry

SECONDARY OUTCOMES:
Day-night rhythm in whole-body energy metabolism (energy expenditure) | measured on day two at 8:00, 13:00, 18:00, 23:00, 04:00
  Energy expenditure (kJ/min) measured by indirect calorimetry
Day-night rhythm in whole-body energy metabolism (glucose oxidation) | measured on day two at 8:00, 13:00, 18:00, 23:00, 04:00
  glucose oxidation (g/min) measured by indirect calorimetry
Day-night rhythm in whole-body energy metabolism (fat oxidation) | measured on day two at 8:00, 13:00, 18:00, 23:00, 04:00
  fat oxidation (g/min) measured by indirect calorimetry
Day-night rhythm in muscle protein levels of markers involved in molecular clock and mitochondrial metabolism. | measured on day two at 8:00, 13:00, 18:00, 23:00, 04:00
  Quantify protein levels by Western blots
Day-night rhythm in muscle DNA of markers involved in molecular clock and mitochondrial metabolism. | measured on day two at 8:00, 13:00, 18:00, 23:00, 04:00
  Quantify DNA by qPCR
Day-night rhythm in muscle DNA involved in molecular clock and mitochondrial metabolism. | measured on day two at 8:00, 13:00, 18:00, 23:00, 04:00
  Quantify DNA by micro-array
Day-night rhythm in muscle mRNA markers involved in molecular clock and mitochondrial metabolism. | measured on day two at 8:00, 13:00, 18:00, 23:00, 04:00
  Quantify mRNA levels by micro array
Day-night rhythm of markers of normal day-night rhythm (cortisol) | measured on day two, every two hours for 24 hours beginning at 08:00
  Blood cortisol levels
Day-night rhythm of in markers of normal day-night rhythm (core body temperature) | measured continuously for 24 hours on day two
  Core body temperature measured by an ingested telemetric pill.
Day-night rhythm of in markers of normal day-night rhythm (melatonin) | measured on day two, every two hours for 24 hours beginning at 08:00
  Blood melatonin levels.
Day-night rhythm in serum glucose | measured on day two, every two hours for 24 hours beginning at 08:00
  Serum glucose levels determined from venous blood draws
Day-night rhythm in serum insulin | measured on day two, every two hours for 24 hours beginning at 08:00
  Serum insulin levels determined from venous blood draws
Day-night rhythm in serum free fatty acids (FFA) | measured on day two, every two hours for 24 hours beginning at 08:00
  Serum FFA levels determined from venous blood draws
Day-night rhythm in serum triglycerides | measured on day two, every two hours for 24 hours beginning at 08:00
  Serum triglyceride levels determined from venous blood draws
Day-night rhythm in serum cholesterol | measured on day two, every two hours for 24 hours beginning at 08:00
  Serum cholesterol levels determined from venous blood draws
Change in energy status of the heart between morning and evening | Measured on first study day 5:30 PM (duration 45 minutes), second study day 7:30 AM (duration 45 minutes)
  variation in phosphorus metabolites measured by Magnetic Resonance Imaging and - Spectroscopy (MRI/MRS)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schrauwen, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wefers J, Connell NJ, Fealy CE, Andriessen C, de Wit V, van Moorsel D, Moonen-Kornips E, Jorgensen JA, Hesselink MKC, Havekes B, Hoeks J, Schrauwen P. Day-night rhythm of skeletal muscle metabolism is disturbed in older, metabolically compromised individuals. Mol Metab. 2020 Nov;41:101050. doi: 10.1016/j.molmet.2020.101050. Epub 2020 Jul 11. PMID 32659272